CLINICAL TRIAL: NCT02466438
Title: Safety and Pharmacokinetics of Piperacillin-Tazobactam Extended Infusions in Infants and Children
Brief Title: Safety and Pharmacokinetics of Piperacillin-tazobactam Extended Infusion in Infants and Children (PIP-TAZO)
Acronym: PIP-TAZO
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Julie Autmizguine, MD, MHS, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUSJ-4131
Record Dates: First submitted 2015-06-02; First posted 2015-06-09 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Infection
Keywords: Antibiotics; Piperacillin-tazobactam; Resistant bacteria
MeSH Terms: conditions — Infections | interventions — Piperacillin, Tazobactam Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Piperacillin-tazobactam (Experimental): Piperacillin-tazobactam administration (fixed combination, ratio piperacillin:tazobactam = 8:1).
  Recruitment stratified by age group and pediatric populations to ensure good representation of those subgroups. Maximum dose: 16g/day. Treatment duration: up to 14 days depending to the treating physician.
  Patients with Normal Renal function:
  * Pediatric and surgery units: 2-5 months (7); 6-11 months (7); 12-23 months (7); 2-6 years (16)
  * Pediatric intensive care unit (PICU): 2-5 months (7); 6-11 months (7); 12-23 months (7); 2-6 years (16)
  * Haematology-oncology unit: 2-5 months (7); 6-11 months (7); 12-23 months (7); 2-6 years (16)
  Patients with Acute Kidney injury:
  * Pediatric and surgery units: 2 months-6 years (10)
  * PICU: 2 months-6 years (10)
  * Haematology-oncology unit: 2 months-6 years (10)
  Interventions: Drug: Piperacillin-tazobactam

INTERVENTIONS:
Drug: Piperacillin-tazobactam — * Normal renal function receiving new optimized piperacillin-tazobactam dosing regimen per age, dosing (mg/kg), duration of infusion
    * Age (2-5 months): 80 mg/kg/dose of medication every 8 hours for 4 hours
    * Age (≥6 months-6y): 130 mg/kg/dose of medication every 8 hours for 4 hours
  * Acute Kidney injury : Dosing as prescribed by treating physician
  Other Names: Piperacillin-tazobactam combination product; Tazocin

SUMMARY:
Severe infection is one of the main causes of disease in hospitalized children and can be deadly. With the lack of novel antibiotics approved in children and the emergence of drug resistant bacteria, there is a critical need to optimize dosing of existing antibiotics. Piperacillin-tazobactam is an antibiotic frequently used for treatment of severe infection in children in Canadian hospitals. To optimize this antibiotic's efficacy despite the rise of antibiotic resistance, alternative dosing strategy is commonly used in adults, which consists of prolonging the time during which the drug is infused (4 hours instead of 30 min). Children clear piperacillin-tazobactam from their bodies at a slower rate than adults, consequently extended-infusion strategy cannot be directly extrapolated from adult to children. We believe that younger children need piperacillin-tazobactam infusions that are shorter compared to adults to achieve appropriate concentrations.

DETAILED DESCRIPTION:
This is a prospective, open-label Pharmacokinetics and safety study of piperacillin-tazobactam in children 2 months-6y of age.

Overall goal: To establish extended-infusion piperacillin-tazobactam dosing recommendations in infants and young children with normal renal function, for the treatment of sepsis due to resistant organisms. Dosing recommendations will be provided according to different levels of antibiotic resistance (MIC). We aim to establish the age threshold below which extended infusion does not provide additional therapeutic benefit because of immature renal function. We also aim to describe the PK of piperacillin-tazobactam standard dosing in children with acute kidney injury.

Study population #1: Normal Renal Function:

Evaluate the PK of piperacillin-tazobactam extended infusion in children 2 months-6y with normal renal function.

Hypothesis 1.1 : Population clearance of piperacillin will be 20% lower in infants 2-5 months compared with infants 6-23 months and will reach adult values at 2 years of age.

Hypothesis 1.2: Alternative dosing strategy used in this clinical trial will achieve pharmacodynamics (PD) target (50% fT > MIC) for minimum inhibitory concentration (MIC) up to 16 mg/L in 90% of infants and children 2 months-6y.

Study Population #2: Acute Kidney Injury:

Describe the PK of piperacillin-tazobactam in children with kidney injury, using the standard dosing.

Hypothesis 2.1: Population clearance of piperacillin will be 15% lower in infants with acute kidney injury but normal glomerular filtration rate (GFR). Clearance will increase as GFR decreases.

Screening:

Infants and children will be screened using a pharmacy software application available in our institution, displaying a list of all subjects meeting inclusion criteria in real time. Recruitment will take place in units where children receive piperacillin-tazobactam.

Enrollment/Baseline: Baseline/Pre-Dose Assessment:

After it has been determined that the participant satisfies all inclusion and no exclusion criteria and after the parent or legal guardian has signed the informed consent form, subjects will be assigned a study number and the following evaluations will be recorded in the clinical research form:

1. Participant demographics including gender, date of birth, chronologic age, corrected age if <1 year of age and born <37 weeks of gestational age, race, birth weight if <1 year of age, and weight at time of consent.
2. Active clinical diagnoses
3. Concomitant medications taken in 72 hours prior to first dose of piperacillin-tazobactam or during treatment with piperacillin-tazobactam
4. Laboratory and microbiologic determinations within 72 hours prior to first dose of piperacillin-tazobactam
5. Microbiological results of sterile body fluids (blood, cerebrospinal fluid (CSF), urine obtained by catheterization or supra-pubic tap), within 72 hours prior to the first dose of study drug

Assessments/Procedures (Day 1 to Day 14): The following assessments will be conducted each day while the patient is on study

1. Study medication administration: The date and time, amount, infusion duration and site of administration of each dose will be recorded. Day 1 will be day of first dose of study drug.
2. PK samples collection: date and time of sample collection, total blood volume collected.
3. Laboratory determinations on each day of PK sample collection
4. Microbiological results of sterile body fluids (blood, CSF, urine obtained by catheterization or supra-pubic tap)
5. Concomitant medications
6. AEs

Follow-up (Day 15 to 17 or End of Therapy): The following assessments will be conducted at end of therapy:

1. Laboratory determinations on the last day of study drug, or within 72h after the last study dose
2. AEs up to 72h after the last study dose

Laboratory Determinations:

Any labs obtained per standard of care may be recorded while the patient is on study at the following timeline: 1) within 72 hours prior to the first dose of study medication 2) within 72h of PK sample collection 3) on Day 14 of therapy (or end of therapy, whichever comes first), or within 72h hours of last study dose will be recorded. If multiple values for a laboratory are obtained in the 72 hours prior to first dose, record the value closest to enrollment.

1. Any hematology values including hemoglobin, hematocrit, white blood cell count, platelet count, and differential.
2. Any serum chemistry values including blood urea nitrogen (BUN), serum creatinine, potassium, sodium, Aspartate transaminase (AST), Alanine transaminase (ALT), albumin.
3. Given that renal function is the main determinant of piperacillin-tazobactam clearance, serum creatinine will be obtained prior to the first study dose, even if not done per standard of care.

Microbiological Determinations:

All results for any cultures obtained of sterile body fluids (blood, CSF, urine obtained by catheterization or supra-pubic tap) from 72 hours prior to first piperacillin-tazobactam dose through the final dose of piperacillin-tazobactam or Day 14 of therapy (whichever comes first) will be recorded in the case report form (CRF).

Special Assays or Procedures: Pharmacokinetics (PK) Samples:

During study treatment, 4 plasma PK samples (200 µL of whole blood/sample) per subject will be collected using an opportunistic approach; PK samples can be collected after any dose of study drug because PK of piperacillin is linear. PK samples will be obtained at the same time as laboratory tests collected per routine medical.

Specimen Preparation, Handling, and Shipping:

PK samples will be collected in ethylenediamine-tetra-acetic acid (EDTA) microcontainers and processed immediately or placed on ice until processing. Samples will be identified using preprinted labels with the protocol number. Plasma will be separated via centrifugation (3000g for 10 minutes at 4°C), manually aspirated and transferred to polypropylene tubes. Plasma samples will be frozen at -80°C freezer until analysis.

Once enrollment and sample collection are completed, PK samples will be shipped on dry ice to a central laboratory where piperacillin and tazobactam plasma concentrations will be measured using a validated bioanalytical assay.

ELIGIBILITY:
Study population #1: Normal renal function

Inclusion Criteria:

* Children 2 months - 6 years of age*
* Piperacillin-tazobactam indicated per standard of care
* Informed consent

Exclusion Criteria:

* Insufficient venous access to allow extended infusion
* History of anaphylaxis to β-lactams
* Supported with extracorporeal membrane oxygenation (ECMO)
* On renal replacement therapy
* Cystic fibrosis
* Acute Kidney injury
* Chronic renal insufficiency defined as defined as a glomerular filtration rate of 10-60 mL/min/1.73 m2

Study population #2: Acute Kidney injury

Inclusion Criteria:

* Children 2 months - 6 years of age
* Piperacillin-tazobactam indicated per standard of care
* Informed consent
* Acute Kidney injury defined as the following:

  * Doubling of serum creatinine according to upper limit of normal for age and gender or
  * Doubling of baseline serum creatinine (defined as the creatinine level at admission, if the value is within normal limit for age and gender) We wil use the smaller value of these 2 definitions to diagnose acute kidney injury in a given subject.

Exclusion Criteria:

* History of anaphylaxis to β-lactams
* Supported with extracorporeal membrane oxygenation (ECMO)
* On renal replacement therapy
* Cystic fibrosis
* Chronic renal insufficiency defined as defined as a glomerular filtration rate of 10-60 mL/min/1.73 m2

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 141 (Estimated)
Dates: Start 2016-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Clearance (CL) for piperacillin and tazobactam | up to 14 days
  Treatment days 1-14 followed by a safety observation period of 3 days after the last study dose.
Proportion of subjects who achieve Pharmacodynamic target (at least 50% of free plasma piperacillin concentration above the MIC [50% fT > MIC]) | up to 14 days
  Treatment days 1-14 followed by a safety observation period of 3 days after the last study dose.
Evaluation of Volume of distribution (V) for piperacillin and tazobactam | up to 14 days
  Treatment days 1-14 followed by a safety observation period of 3 days after the last study dose.

SECONDARY OUTCOMES:
Proportion of subjects experiencing adverse events (AEs) | up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Julie Autmizguine, MD, MHS, Principal Investigator — St. Justine's Hospital
Locations (1):
- St. Justine's Hospital, Montreal, Quebec, Canada